CLINICAL TRIAL: NCT01432171
Title: Randomized, Double-Blind, Placebo-Controlled Trial of Lacosamide for Seizure Prophylaxis in Patients With High-Grade Gliomas
Brief Title: Lacosamide in Preventing Seizures in Participants With Malignant Glioma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BTTC11-01; NCI-2018-01854 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); BTTC11-01 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2011-09-08; First posted 2011-09-12 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Malignant Glioma
MeSH Terms: conditions — Glioma | interventions — Lacosamide; 2-(acetylamino)-3-methoxy-N-(phenylmethyl)-, (2R)-

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (lacosamide) (Experimental): Participants receive lacosamide PO BID for up to 1 year. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Lacosamide
- Arm II (placebo) (Placebo Comparator): Participants receive a placebo PO BID for up to 1 year. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lacosamide — Given PO
  Other Names: ADD 234037; Erlosamide; Harkoseride; SPM 927; Vimpat
  Arms: Arm I (lacosamide)
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (placebo)

SUMMARY:
This trial studies how well lacosamide works in preventing seizures in participants with malignant glioma. Anti-seizure drugs, such as lacosamide, may decrease abnormal electrical activity in the brain that plays a role in developing seizures.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if prophylactic administration of Lacosamide reduces the risk of seizures in patients with high-grade glioma (HGG).

SECONDARY OBJECTIVES:

I. To determine the one-year risk of first seizure in this patient population. II. To evaluate patient reported symptoms.

EXPLORATORY OBJECTIVES:

I. To investigate clinical and electroencephalographic predictors of seizures in this patient population.

II. To evaluate the occurrence of symptoms and correlate to seizure activity as well as tolerance to treatment using the MD Anderson Symptom Inventory-Brain Tumor Module (MDASI-BT) self-reporting tool.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I (LACOSAMIDE): Participants receive lacosamide orally (PO) twice a day (BID) for up to 1 year. Treatment continues in the absence of disease progression or unacceptable toxicity.

ARM II (PLACEBO): Participants receive a placebo PO BID for up to 1 year. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up every 3 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed supratentorial high-grade glioma will be eligible for this protocol.
* All patients must sign an informed consent indicating that they are aware of the investigational nature of this study.
* Patients must have signed an authorization for the release of their protected health information.
* Patients must have a Karnofsky performance status of >= 60.
* Women of childbearing potential must have a negative beta-human chorionic gonadotropin (HCG) pregnancy test documented within 2 weeks prior to registration.
* In the opinion of the treating investigator, patients must have adequate cognitive abilities to complete the neurocognitive components of the study.
* Patients must be able to safely swallow pills.
* Patients must agree to practice adequate contraception.
* Patients must be registered on study within 16 weeks after the surgical procedure that established the diagnosis of high grade glioma.

Exclusion Criteria:

* Patients must not have any significant medical or psychiatric illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy.
* Patients must not have serious intercurrent medical illness. Serious, active co-morbidity, defined as follows: a) Unstable angina and/or congestive heart failure requiring hospitalization within the last 12 months. b) Transmural myocardial infarction within the last 6 months. c) Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration. d) Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration. e) Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol. f) Acquired immune deficiency syndrome (AIDS) based upon current Centers for Disease Control (CDC) definition; note, however, that human immunodeficiency virus (HIV) testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive. g) Active connective tissue disorders, such as lupus or scleroderma, that in the opinion of the treating physician may put the patient at high risk for radiation toxicity.
* Patients must not be pregnant or breast feeding. Patients must not be pregnant because lacosamide produced developmental toxicity in rats following administration during pregnancy. There is insufficient information to determine if lacosamide is safe during lactation.
* Patients must not have any disease that will obscure toxicity or dangerously alter drug metabolism.
* Patients must not have a history of heart block or cardiac arrhythmia, including asymptomatic arrhythmias and atrial fibrillation/flutter.
* Patients must not have a prolonged PR interval (defined as > 200 ms).
* Perioperative anticonvulsants should be tapered as indicated in the protocol.
* Patients must not have a history of any type of seizure for at least 10 years prior to registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-07-25 (Actual); Primary Completion 2017-06-20 (Actual); Study Completion 2017-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marta Penas-Prado, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: July 25, 2012 to May 23, 2016. All recruitment done in medical clinical settings.
Groups:
- Lacosamide (Vimpat): Lacosamide orally twice a day, starting dose 50 mg with dose escalation (increased by 100 mg/day weekly) until target dose 200 mg achieved over 4 weeks
- Placebo: Placebo orally twice a day.
Period: Overall Study
Arm/Group | Lacosamide (Vimpat) | Placebo
Started | 18 | 19
Completed | 4 | 8
Not Completed | 14 | 11
Not completed — Death | 1 | 2
Not completed — Lost to Follow-up | 6 | 5
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Noncompliance | 2 | 3
Not completed — Insurance denial trial coverage | 1 | 0
Not completed — Patient moved to palliative care | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Lacosamide: Lacosamide orally twice a day, starting dose 50 mg with dose escalation (increased by 100 mg/day weekly) until target dose 200 mg achieved over 4 weeks
- Total: Total of all reporting groups
Arm/Group | Lacosamide | Placebo | Total
Number analyzed (Participants) | 18 | 19 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 15 | 29
  >=65 years | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (12) | 60 (10) | 57 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 12 | 12 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 18 | 19 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 15 | 18 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 18 | 19 | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Seizures
Description: Number of Participants that had seizure in a randomized, two-arm, parallel groups of post-operative participants with newly-diagnosed high-grade glioma (HGG)
Time Frame: 12 months or first seizure
Measure: Count of Participants; unit: Participants
Arm/Group | Lacosamide | Placebo
Number analyzed (Participants) | 18 | 19
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse event data collected for up to one year treatment period.
Arm/Group | Lacosamide | Placebo
All-Cause Mortality (participants affected / at risk) | 1/18 | 2/19
Serious Adverse Events (participants affected / at risk) | 2/18 | 6/19
Other Adverse Events (participants affected / at risk) | 16/18 | 17/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (N=18) | Placebo (N=19)
headache (Nervous system disorders) | 0 (0) | 1 (1)
confusion (Psychiatric disorders) | 1 (1) | 2 (2)
hallucinations (Psychiatric disorders) | 0 (0) | 1 (1)
memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
gait disturbance (General disorders) | 0 (0) | 1 (1)
lung infection (Infections and infestations) | 0 (0) | 1 (1)
neoplasms benign, malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
platelet count decreased (Investigations) | 0 (0) | 2 (2)
white blood cell count decreased (Investigations) | 0 (0) | 2 (2)
neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
hypotension (Vascular disorders) | 1 (1) | 0 (0)
lethargy (Nervous system disorders) | 1 (1) | 0 (0)
seizure (Nervous system disorders) | 0 (0) | 1 (1)
infection, possible sepsis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (N=18) | Placebo (N=19)
platelet count decreased (Investigations) | 0 (0) | 2 (6)
white blood cell decreased (Investigations) | 0 (0) | 2 (8)
alanine aminiotransferase increased (Investigations) | 0 (0) | 2 (2)
blood bilirubin increased (Investigations) | 0 (0) | 1 (4)
neutrophil count decreased (Investigations) | 0 (0) | 1 (4)
muscle weakness, left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
muscle weakness, right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
eye disorders, other (Eye disorders) | 0 (0) | 1 (2)
constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2)
gastrointestinal disorders, other (Gastrointestinal disorders) | 0 (0) | 2 (2)
fatigue (General disorders) | 2 (3) | 5 (5)
gait disturbance (General disorders) | 1 (2) | 2 (4)
infections and infestations, other (Infections and infestations) | 2 (2) | 1 (1)
neoplasms benigh, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1)
anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
thromboembolic event (Vascular disorders) | 3 (3) | 2 (2)
hypertension (Vascular disorders) | 0 (0) | 2 (3)
surgical and medical procedures (Surgical and medical procedures) | 4 (6) | 0 (0)
alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
dyspnea (Nervous system disorders) | 2 (2) | 0 (0)
dysphasia (Nervous system disorders) | 0 (0) | 2 (2)
headache (Nervous system disorders) | 4 (4) | 5 (5)
memory impairment (Nervous system disorders) | 0 (0) | 2 (2)
seizure (Nervous system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This is a cooperative group protocol. It was not an MDACC protocol. BTTC was administratively located at MDACC. The main PI/Academic PI was located at an outside institution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-05-30): https://cdn.clinicaltrials.gov/large-docs/71/NCT01432171/Prot_SAP_000.pdf